CLINICAL TRIAL: NCT04287166
Title: Feasibility of Remote Early At-risk Diagnosis for Cerebral Palsy in High-risk Infant Follow-up Clinics in The Central Norway Regional Health Authority
Brief Title: Early Remote At-risk Diagnosis for Cerebral Palsy in Follow-up Clinics for High-risk Infants
Acronym: In-Motion
Status: Active, not recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Alesund Hospital (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: REK 62240
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy
Keywords: Diagnosis; Videos; Smartphone app; Movement; Movement disorders; Infants
MeSH Terms: conditions — Cerebral Palsy; Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral Palsy (CP) is the most common motor dysfunction in childhood. Traditionally, diagnosis is set between 12 and 24 months of age. This study will evaluate feasibility of a new screening procedure for early detection of CP in high-risk infants and investigate how such a procedure can be implemented in the Central Norwegian Regional Health Authority (CNRHA).

The most accurate method to detect and predict CP at an early age is the General Movement Assessment (GMA). GMA is based upon expert observations of infant spontaneous movements in a video. In Central-Norway such expertise is today only present at St. Olavs Hospital, Trondheim University Hospital. Video recordings by health personnel and parents will be used in follow-up programs within CNRHA for remote expert based GMA. In addition, machine learning models will be applied for automatic detection of CP.

Early identification of CP will lead to improved function and increased possibility to direct health care resources to the patients who need it most, independent of geographical and expert based constraints.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized at a Neonatal Intensive Care Unit (NICU) within the Central Norway Regional Health Authority that is referred to follow-up in the Specialist Health Services containing a team of minimum a pediatrician and a physiotherapist.
* at high-risk for adverse neurological outcomes as considered by the pediatrician on the basis of clinical judgement (example: serious asphyxia, prematurity, stroke, brain hemorrhage)

Exclusion Criteria:

* Peripheral neuromotor disease e.g. brachial plexus injury
* iatrogenic restricted movements (e.g. cast for clubfoot)

Ages: 0 Months to 2 Months | Sex: All
Age Groups: Child
Study Population: High-risk infants referred to high-risk follow-up at discharge from one of the participating Neonatal Intensive Care Units, are candidates for enrollment. Following review of the inclusion and exclusion criteria, eligible subjects will be invited to participate. All subjects (parents) must give written informed consent prior to any study procedures being carried out.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Scorable video for remote GMA | 1 week
Correlation of computer software data between standard video set-up and handheld smartphone video. | 1 week
Predictability of GMA and computer-based assessment for development of CP | 2 years
Predictability of GMA and computer-based assessment for development of CP | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lise Støylen, Study Director — St Olavs Hospital, Clinic of Clinical Services; Torstein Rø IKOM, Study Director — Norwegian University of Science and Technology, IKOM
Locations (3):
- Norway (3):
  - Department of Pediatrics, Møre and Romsdal Hospital Trust, Ålesund
  - Department of Pediatrics, Nord-Trøndelag Hospital Trust, Levanger
  - Department of Pediatrics, St. Olav's Hospital Trust, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adde L, Aberg KB, Fjortoft T, Grunewaldt KH, Lade R, Osland S, Piegsa F, Sandstrom PG, Stoen R, Storvold GV, Eriksen BH. Implementation of remote general movement assessment using the in-motion instructions in a high-risk norwegian cohort. BMC Pediatr. 2024 Jul 10;24(1):442. doi: 10.1186/s12887-024-04927-4. PMID 38987721